CLINICAL TRIAL: NCT05978414
Title: Functional Relationships Between the Temporomandibular Joint and the Pelvis in Women With Gynecological Diseases of Genital Prolapse and Endometriosis
Brief Title: Functional Links Between the Temporomandibular Joint and the Pelvis in Gynecology
Acronym: TMJ and Pelvis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: University of Life Science in Poznan (Unknown)
Responsible Party: Principal Investigator, Małgorzata Wójcik, PhD PT, principal investigator, research manager, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 305/23
Record Dates: First submitted 2023-06-28; First posted 2023-08-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Prolapse; Female; Endometriosis-related Pain
Keywords: quaity of life; women; prolapse; female; endometriosis-related pain; visceral therapy; temporomandibular joint
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Intervention Model Description: Description of the study group: The study will qualify women, aged from 18 to 60 years old admitted to the Sredz Heart Hospital in Sroda Wielkopolska, gynecology and obstetrics department. The planned study group is 200 women after surgical treatment (100 with prolapse of reproductive organs and 100 with a diagnosis of endometriosis). Both conditions are planned to be randomly divided into: a subgroup undergoing physiotherapy intervention and a subgroup without physiotherapy intervention. Women who do not consent to physiotherapeutic intervention will be included in the control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Women will be randomly assigned to a test and control group according to their disease. The person performing the visceral tests and techniques will not know which group the woman belongs to. The evaluator of the results will not know whether they are the group with or without visceral techniques.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 subgroups with wisceral therapy (Experimental): A group of women with endometriosis and reproductive organ prolapse will be randomly assigned to the intervention will have visceral therapy performed, and the group without the intervention will have a placebo.
  Interventions: Other: Visceral therapy
- 2 subgroups with placebo (without intervention) (Placebo Comparator): The group of women with endometriosis and reproduvtive organ prolapse without the intervention will have a placebo only hands held on the pelvis by a physiotherapist.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Visceral therapy — Visceral therapy will be performed manually by a physiotherapist, a detailed description of the techniques is above. Therapy will be in 2 subgroups with prolapse of the usual genitals and endometriosis.
  Arms: 2 subgroups with wisceral therapy
Other: Placebo — Placebo will be in 2 subgroups that will not have visceral therapy. The placebo will consist of the physiotherapist holding hands on the patient's pelvis.
  Arms: 2 subgroups with placebo (without intervention)

SUMMARY:
1 Recruitment. 2. Collection of written consents for the study. 3. Random assignment to groups with and without intervention. 4. Completion of questionnaires by study participants, postural pattern assessment, temporomandibular joint assessment, and platform assessment.

5. Performance of visceral therapy in the group with intervention, in the group without intervention placebo. Duration 5 weeks, treatment 1x per week at the same time of day and given day e.g. Mondays only.

6. Reassessment as in step 4. 7. Data collection, statistical analyses. 8. Interpretation of results for female participants. 9. Preparation of results for scientific publications.

DETAILED DESCRIPTION:
Methods

After taking a detailed history, patients will be asked to:

1. Completing: the SF-36 quality of life assessment questionnaire and Female Sexual Function Index assessment, and marking on a numerical scale their pain sensations for the temporomandibular joint and for the pelvis, World Health Organization Quality of Life BREF (WHOQOL-BREF).

   The SF-36 questionnaire, FSFI scale, World Health Organization Quality of Life BREF (WHOQOL-BREF) and numerical scale (assessing pain sensations for the temporomandibular joint and pelvic joint), will also be subjected to completion/checking after the completion of manual visceral treatments in groups with physiotherapy intervention for both conditions.
2. Type of postural pattern according to Hall-Wernham-Littlejohn: type I - normal, type II - anterior pelvic tilt, type III - posterior pelvic tilt.

3 Pelvic type assessment: normal, high, low; pelvic type will be assessed in each patient and in groups with physiotherapeutic intervention for both conditions before and after manual visceral treatments.

4. Assessment of mobility in the temporomandibular joints in the sagittal plane CromWell digital caliper, and diagnosis using standardized protocols.

5. Postural assessment on the Posturomed Technomex platform and Podoscope Sensor Medica.

6. 6.Manual visceral treatments The treatments will be performed after the patient is qualified by the obstetrician-gynecologist specialist.

7. After performing techniques and placebo in both groups, filling out questionnaires again, measuring on the platform, pattern posture..

8. Statistical analysis: upon completion of the study, the collected quantitative and qualitative data will be subjected to statistical analysis. The choice of statistical tools will depend on the obtained probability distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Written consent to participate in the study.
2. Female patients after surgical treatment with prolapse of reproductive organs and diagnosed endometriosis.

Exclusion Criteria:

1. No written consent to participate in the study.
2. Cancer.
3. Injury to the temporomandibular joint and pelvis.
4. Fibromyalgia.
5. Rheumatic diseases.
6. At each stage of the experiment if the patient decides that she does not want to participate she is excluded.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The study will include women because diseases like endometriosis and genital prolapse are diseases of women.
Enrollment: 200 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
NRS | Time point one: before starting visceral therapy and placebo, 1 st week
  Each patient will mark on the NRS scale the sensation of pain before the tests. Scale of 1-10, the higher the value the greater the pain experience.
platforms | Time point one: before starting visceral therapy and placebo,1 st week
  Each patient will have a postural stability assessment prior to testing.No platform manufacturer provides standards. The platform is equipped with sensors - it collects the force of the feet and gives how the center of gravity is located, that is, the front-back, side-to-side tilts are given.
postural pattern by Halla-Wernhama-Littlejohna | Time point one: before starting visceral therapy and placeb1 st weeko,
  Before the test, each patient will have a postural pattern assessment. Evaluating the pattern of type 1 anterior tilt of the body, type 2 normal, type 3 posterior tilt.
pelvic type assessment | Time point one: before starting visceral therapy and placebo,1 st week
  Before the test, each patient will have a pelvic type assessment. High-assimilated type: hip plates above the L5 segment: overloaded type: hip plates below the L4 segment; normal type: hip plates at the level of the L4-L5 segment.
CromWell (measurement of oral dilation) | Time point one: before starting visceral therapy and placebo,1 st week
  Before the test, each patient will have their mouth opening measured with an electronic caliper.There are no standards given, it is a measurement of the dilation of the mouth.
standarised questonarie by Kulesa-Morawiecka et al. | Time point one: before starting visceral therapy and placebo,1 st week
  Each patient will complete a questionnaire on the evaluation of the temporomandibular joint. Scale of 0-10 points, 0 - means no strength of head and neck muscles, 10 - means strong tension of head and neck muscles.
According to the Polish version of the questionnaire, the highest point value, i.e. 171, indicates the lowest rank in the quality of life assessment, while the lowest point value indicates the highest level of quality of life. | Time point one: before starting visceral therapy and placebo,1 st week
  Each patient will complete a questionnaire on the evaluation of quality of life.Assessment: physical functioning, limitations due to physical health, pain perception, general sense of health, vitality, social functioning, emotional functioning and mental health.
Female Sexual Function Index. Score: a value of 26 points or less indicates the presence of significantly clinical sexual dysfunction. | Time point one: before starting visceral therapy and placebo,1 st week
  Each patient will complete a questionnaire.
visceral techniques and placebo | 1 st week, 2nd week, 3rd week,4th week, 5 week
  The intervention group will have visceral therapy performed. The group without intervention will only have their hands held on the pelvis.

SECONDARY OUTCOMES:
NRS | Time point two: after visceral therapy and placebo, 5th week
  After 5 weeks, each patient will mark on the pain sensation scale. Scale of 1-10, the higher the value the greater the pain experience.
platforms | Time point two: after visceral therapy and placebo, 5th week
  After 5 weeks, each patient will have a postural stability assessment. No platform manufacturer provides standards. The platform is equipped with sensors - it collects the force of the feet and gives how the center of gravity is located, that is, the front-back, side-to-side tilts are given.
postural pattern by Halla-Wernhama-Littlejohna | Time point two: after visceral therapy and placebo, 5th week
  After 5 weeks, each patient will have a posture pattern assessment. Evaluating the pattern of type 1 anterior tilt of the body, type 2 normal, type 3 posterior tilt.
pelvic type assessment | Time point two: after visceral therapy and placebo,5 th week
  After 5 weeks, each patient will have a pelvic type assessment.High-assimilated type: hip plates above the L5 segment: overloaded type: hip plates below the L4 segment; normal type: hip plates at the level of the L4-L5 segment.
CromWell (measurement of oral dilation) | Time point two: after visceral therapy and placebo, 5th week
  After 5 weeks, each patient will have an evaluation of oral dilation with an electronic caliper.There are no standards given, it is a measurement of the dilation of the mouth.
standarised questonarie by Kulesa-Morawiecka et al. | Time point two: after visceral therapy and placebo, 5th week
  After 5 weeks, each patient will complete a temporomandibular joint evaluation questionnaire.Scale of 0-10 points, 0 - means no strength of head and neck muscles, 10 - means strong tension of head and neck muscles.
According to the Polish version of the questionnaire, the highest point value, i.e. 171, indicates the lowest rank in the quality of life assessment, while the lowest point value indicates the highest level of quality of life. | Time point two: after visceral therapy and placebo, 5th week
  After 5 weeks, each patient will complete a quality of life questionnaire. Assessment: physical functioning, limitations due to physical health, pain perception, general sense of health, vitality, social functioning, emotional functioning and mental health.
Female Sexual Function Index. Score: a value of 26 points or less indicates the presence of significantly clinical sexual dysfunction. | Time point two: after visceral therapy and placebo, 5th week
  After 5 weeks, each patient will complete a sexual satisfaction questionnaire
World Health Organization Quality of Life BREF (WHOQOL-BREF) | Time point two: after visceral therapy and placebo, 5th week
  After 5 weeks, each patient will complete a sexual satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Physical Education, Poznan, Poland